CLINICAL TRIAL: NCT01844206
Title: Two Dose Epidural Morphine for Post-cesarean Analgesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment of subjects
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Allison Lee, Assistant Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAL3857
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Pain; Morphine Adverse Reaction
Keywords: Post-cesarean analgesia; Second dose of epidural morphine after surgery; Post-operative analgesia; Self-administered epidural morphine; Pain management after cesarean
MeSH Terms: conditions — Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural Morphine (Active Comparator): Group receiving 3mg epidural morphine, 24 hours after the initial dose
  Interventions: Drug: Epidural Morphine
- Epidural Saline (Placebo Comparator): Group receiving epidural saline 6ml, 24 hours after receiving epidural morphine 3mg.
  Interventions: Drug: Epidural Saline

INTERVENTIONS:
Drug: Epidural Morphine — Patients will be given 3mg epidural morphine, 24 hours after the initial dose.
  Other Names: DepoDur
  Arms: Epidural Morphine
Drug: Epidural Saline — Patients will be given epidural saline 6ml, 24 hours after receiving epidural morphine 3 mg.
  Other Names: Sodium Chloride Solution
  Arms: Epidural Saline

SUMMARY:
The investigators aim to assess the analgesic effect of a two-dose epidural morphine regimen for 2nd day post-cesarean pain, as part of a multimodal analgesia regimen, which includes scheduled Nonsteroidal anti-inflammatory drugs (NSAIDs). The investigators hypothesize that administration of a second dose of epidural morphine 3 mg, 24 hours after an initial intraoperative dose, will provide superior post-cesarean analgesia during the 2nd 24 hours after surgery, compared to a single epidural morphine dose regimen. The primary outcome will be the amount of intravenous morphine patients self-administer during the 2nd 24 hours post-surgery.

DETAILED DESCRIPTION:
This will be a randomized, double-blinded placebo-controlled study. In this study, women who underwent cesarean section with epidural anesthesia will receive 3 mg of epidural morphine intraoperatively, and have the epidural catheter left in place. Patients will be randomized to receive either epidural saline or epidural morphine 3 mg at 18 - 24 hours after the first dose of epidural morphine, following which the epidural catheter will be removed. It is standard of care at our institution for women undergoing cesarean section with epidural anesthesia to receive epidural morphine 3 mg. What is not typically carried out is to give a second dose of epidural morphine 3mg.

The randomization will be carried out by a computerized block randomization table; the proportion for the 2 groups will be 1:1. The primary outcome will be the amount of intravenous morphine patients self-administer in the second 24 hours after surgery. Secondary outcomes will include pain scores every 6 hours, satisfaction with analgesia, side effects (itching, nausea/vomiting).

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean section under epidural anesthesia.

Exclusion Criteria:

* Emergent cesarean section
* Coagulopathy
* Failed epidural anesthesia or patchy block
* General anesthesia
* Use of epidural chloroprocaine
* Allergy or contraindication to Non-steroidal anti-inflammatory drug (NSAIDs)
* Severe opioid side effects
* History of chronic opioid use
* History of chronic pain
* History of obstructive sleep apnea
* Morbid obesity (Body Mass Index (BMI)>45 kg/m2)
* Height under 4' 10" (147 cm)
* Documented dural puncture by the epidural (Tuohy) needle
* Preeclampsia
* Other significant medical disease (American Society of Anesthesiologists (ASA) 3 or more).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lee, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Background] Zakowski MI, Ramanathan S, Turndorf H. A two-dose epidural morphine regimen in cesarean section patients: pharmacokinetic profile. Acta Anaesthesiol Scand. 1993 Aug;37(6):584-9. doi: 10.1111/j.1399-6576.1993.tb03769.x. PMID 8213024
- [Background] Palmer CM, Nogami WM, Van Maren G, Alves DM. Postcesarean epidural morphine: a dose-response study. Anesth Analg. 2000 Apr;90(4):887-91. doi: 10.1097/00000539-200004000-00021. PMID 10735794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epidural Morphine | Epidural Saline
Started | 2 | 3
Completed | 2 | 2 (One patient requested that epidural catheter be removed during the first post-operative day.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Morphine | Epidural Saline | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Average Amount of Intravenous Morphine Patients Self-administered in the Second 24 Hours Post-surgery
Description: The primary outcome of this study is the amount (mg) of morphine self-administered by PCA pump during the second 24 hours after surgery. This will be compared by unpaired t-test for two groups.
Time Frame: Up to 48 hours post-operatively
Population: Data could not be summarized to include in the data table because only 5 out of 140 subjects were enrolled prior to study termination, and no data analysis was carried out. As instructed, we are specifying zero ("0") for the Number of Participants Analyzed in each Arm/Group and leaving the data fields blank.
Arm/Group | Epidural Morphine | Epidural Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 hours post-surgery
Description: Women undergoing cesarean section under epidural anesthesia virtually always receive epidural morphine for post-operative analgesia. The 5 women did not experience any unexpected/reportable serious or non-serious adverse effects from the epidural morphine after cesarean section.
Arm/Group | Epidural Morphine | Epidural Saline
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No